CLINICAL TRIAL: NCT00956176
Title: Intravesical Cidofovir Instillation in HSCT Recipients With Hemorrhagic Cystitis: A Single Dose Pharmacokinetic Study
Brief Title: Cidofovir Instillation in Hematopoietic Stem Cell Transplant (HSCT) Recipients With Hemorrhagic Cystitis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0040
Record Dates: First submitted 2009-08-07; First posted 2009-08-11 (Estimated); Last update posted 2019-05-14 (Actual); Status verified 2019-05

CONDITIONS: Cystitis; Bladder Diseases
Keywords: Cidofovir; Vistide; Adenovirus; BK virus infections; HSCT; Hemorrhagic Cystitis; Foley catheter; Viral infection; Bladder instillation; Intravesical; Transurethral catheter; Transplantation
MeSH Terms: conditions — Cystitis; Urinary Bladder Diseases; Adenoviridae Infections; Cystitis, Hemorrhagic; Virus Diseases | interventions — Cidofovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cidofovir (Experimental)
  Interventions: Drug: Cidofovir

INTERVENTIONS:
Drug: Cidofovir — Single dose of 5 mg/kg administered in 100 ml of normal saline solution through a foley catheter to bladder. The catheter will be clamped for 2 hours to keep the drug in bladder.
  Other Names: Vistide

SUMMARY:
The goal of this clinical research study is to learn how the body absorbs and processes 1 dose of cidofovir that is given directly into the bladder, in patients with a viral infection that is causing bleeding from the bladder.

The safety of this drug dose and the investigational way it is given (directly into the bladder) will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

Cidofovir is designed to fight CMV (a viral infection) by blocking the CMV cells from dividing.

Cidofovir is commonly given by injection. For research purposes, in this study it will be given directly into the bladder through a foley catheter. This is one of the first studies where cidofovir is being given this way in humans.

Study Drug Administration:

If you are found to be eligible to take part in this study, on Day 1, Cidofovir will be put into your bladder through your foley catheter. The catheter will be clamped for 2 hours to keep the drug in your bladder. After 2 hours, the catheter will be unclamped. If you were receiving bladder irrigation as therapy for your hemorrhagic cystitis, this will be restarted.

Study Tests on Day 1:

On the day you receive cidofovir, blood (about 2 teaspoons) will be drawn 6 times. The first blood draw will occur before the cidofovir dose, and the last blood draw will occur 24 hours (+/- 1 hour) after the start of the dose. This blood will be used for pharmacokinetic (PK) and pharmacodynamic (PD) testing. PK testing measures the amount of study drug in the body at different time points. PD testing is used to look at how the level of study drug in your body may affect the disease.

Viral Load Testing:

During this study, extra urine and leftover blood to be collected and used for research to test for certain viruses. These viruses include the type of infection you had when joining this study, as well as cytomegalovirus (CMV) and another type of herpes virus.

The urine samples will be collected before the cidofovir dose on Day 1, after the cidofovir dose on Day 1, and again on Day 4.

Any blood left over from Day 1 testing will also be used for viral load testing.

It is possible that these urine and/or blood samples will be sent to an outside lab to perform this testing. If that occurs, your name and any personal identifying information will be coded before the samples are sent. Coding the samples is designed to protect your privacy.

Follow-Up Tests:

Blood (about 2 teaspoons) will be drawn for routine tests 2 times during the week after your cidofovir dose.

On Day 7 (+/- 2 days), you will be checked for any side effects that could be related to the study drug.

In addition, on Day 14 (+/- 2 days), blood samples will be drawn for PK testing, urine will be collected for routine tests, and your safety data will be recorded.

One final follow-up visit will take place on Day 30 (+/- 2 days). During this visit, the study staff will record any serious side effects you may be experiencing.

Length of Study Participation:

Your active study participation will be over after the Day 7 follow-up visit (+/- 2 days). If you experienced a side effect, however, the study staff will continue checking your medical records until the side effect becomes stable or gets better.

This is an investigational study. Cidofovir given by injection is commercially available and FDA approved to treat CMV in patients with HIV. It is investigational to give cidofovir directly into the bladder of patients who have a viral infection causing bleeding in the bladder.

Up to 6 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Polyoma BK or adenovirus viruria has been established either by positive urine cytology or by PCR for BK virus or by positive urine and/or blood culture for adenovirus
2. The patient has either gross hematuria and/or passes blood clots
3. Signed informed consent form
4. Hospitalized patients with a Foley catheter
5. Women of childbearing potential must agree to use 2 acceptable methods of birth control (e. g., abstinence, IUD, or barrier method), during the study period and one for a period of 2 months afterward. At least one of the methods must be a barrier method. Males must also agree to use acceptable method of birth control (barrier method) during the study period and for 2 months afterward.

Exclusion Criteria:

1. Serum creatinine >1.5 mg/dl and/or calculated creatinine clearance < 55 ml/min using the Cockcroft-Gault Creatinine Clearance formula (CrCl). CrCl = {(140-Age) x Weight (kgs) x 0.85 (if female)}/ {72x Serum Creatinine (mg/dl)}
2. Urine protein > 100 mg/dl (equivalent to > 2+ proteinuria)
3. Age less than 18 years
4. Prior therapy with formalin or carboprost 1 mg % administered intravesically
5. Hypersensitivity to cidofovir, probenecid or sulfa-containing medications
6. Have received prior cidofovir therapy within 2 weeks.
7. Prior enrollment in the study
8. Women who are pregnant or breast-feeding
9. Evidence of end-organ adenoviral infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Systemic Absorption of Cidofovir via bladder instillation | Blood collected pre-instillation, 1 hour, 2 hours, 4 hours and 14 hours after instillation.

CONTACTS AND LOCATIONS:
Overall Officials: Roy F. Chemaly, MD, MPH, MBA, Principal Investigator — UT MD Anderson Cancer Center

REFERENCES:
- See also: UT MD Anderson Cancer Center — http://www.mdanderson.org